CLINICAL TRIAL: NCT00043888
Title: A Phase IIIb/IV, Randomized, Open Label, Multicenter, Pilot Trial to Explore the Safety and Tolerability of GW433908 +/- Ritonavir (1400mg Twice Daily or 700mg/100mg Twice Daily) When Used in Combination With a Zidovudine-containing Regimen (TRIZIVIR or COMBIVIR Twice Daily) Over a 24 Week Period in Antiretroviral Therapy Naive HIV-1 Infected Subjects.
Brief Title: Study to Explore Safety And Tolerability of Fosamprenavir With or Without Ritonavir in Combination With TRIZIVIR or COMBIVIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZL30006
Record Dates: First submitted 2002-08-14; First posted 2002-08-19 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: fosamprenavir; ritonavir; COMBIVIR; TRIZIVIR; abacavir; lamivudine; zidovudine; HIV; protease inhibitors
MeSH Terms: conditions — HIV Infections | interventions — fosamprenavir; lamivudine, zidovudine drug combination; Ritonavir; abacavir, lamivudine, and zidovudine drug combination

INTERVENTIONS:
Drug: fosamprenavir
Drug: COMBIVIR
Drug: ritonavir
Drug: TRIZIVIR

SUMMARY:
Antiretroviral Therapy (ART) naive subjects will be enrolled in this clinical research study to test the safety and tolerability of fosamprenavir with or without ritonavir in combination TRIZIVIR and COMBIVIR. Subjects will receive 24 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Lab result for Screening viral load (HIV-1 RNA) greater than or equal to 1,000 copies per mL.
* Lab result for Screening CD4 cell count greater than or equal to 100 cells per microliter.
* Antiretroviral therapy naive (no prior therapy allowed).
* Male or female 13 years of age or older (or 18 years of age or older according to local requirements).
* Female subjects must be of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including women who are post-menopausal) or of child-bearing potential with a negative blood pregnancy test at screen and who agree to use a proven barrier method of contraception (e.g. spermicide plus condom) during the study period. Hormonal contraceptives will not be considered sufficient forms of contraception for this study. All subjects participating in this study should be counselled on the practice of safe or safer sex.
* Able to understand and provide written informed consent to participate in this trial. Parental or guardian consent must also be obtained for subjects under the age of 18 years.

Exclusion Criteria:

* Prior history of having received antiretroviral therapy.
* An active HIV Associated Disease (Center for Disease Control Category C) within 28 days of study drug administration.
* Any sudden onset or sharp rise in a laboratory abnormality (including abnormally high laboratory values) at Screening that causes the investigator to have the opinion that the subject should not participate in the study of an investigational compound.
* Subjects with a laboratory result for estimated creatinine clearance less than 40 ml per minute within 28 days of study drug administration.
* Laboratory result for serum aminotransferase (AST, ALT) levels elevated greater than five to ten times (or more) the upper limit of the normal range within 28 days prior to study drug administration.
* Pregnant or lactating women.
* History of clinically relevant pancreatitis or hepatitis within 6 months of study drug administration.
* Presence of any serious medical condition (e.g., diabetes, cardiac dysfunction, hepatitis) which, in the opinion of the investigator, might compromise the safety of the subject.
* Presence of a malabsorption syndrome or other gastrointestinal dysfunction which might interfere with drug absorption or render the subject unable to take oral medication.
* History of a drug or other allergy which, in the opinion of the investigator, contraindicates the subject's participation in the study.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days of study drug administration or anticipated need for such treatment during the study.
* Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 28 days of study drug administration.
* Treatment with any HIV vaccine within 3 months of study drug administration.
* Treatment with other selected medications within 28 days prior to receiving study medication or the anticipated need during the study.
* Current alcohol or illicit drug use which, in the opinion of the investigator, may interfere with the subject's ability to comply with the requirements of the study. Note: Subjects stabilized on methadone can be considered for participation.
* Treatment with other investigational drugs or therapies within 28 days prior to Day 1, or an anticipated need for such treatment during the study. Treatments available through a Treatment IND or other expanded-access mechanism will be evaluated on a case-by-case basis.
* Other inclusion or exclusion criteria to be determined by the investigator and sponsor of the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2002-01; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
To assess the overall short term tolerance of the regimens under investigation

SECONDARY OUTCOMES:
Nature and incidence of laboratory abnormality; impact/burden of adverse events to subjects; plasma zidovudine (ZDV)pharmacokinetic parameters; change from baseline in plasma HIV-1 RNA levels over time.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD, Study Director — GlaxoSmithKline
Locations (15):
- United States (11):
  - GSK Clinical Trials Call Center, Little Rock, Arkansas
  - GSK Clinical Trials Call Center, Long Beach, California
  - GSK Clinical Trials Call Center, Newport Beach, California
  - GSK Clinical Trials Call Center, San Diego, California
  - GSK Clinical Trials Call Center, Denver, Colorado
  - GSK Clinical Trials Call Center, Washington D.C., District of Columbia
  - GSK Clinical Trials Call Center, Altamonte Springs, Florida
  - GSK Clinical Trials Call Center, Fort Lauderdale, Florida
  - GSK Clinical Trials Call Center, Atlanta, Georgia
  - GSK Clinical Trials Call Center, Greenville, North Carolina
  - GSK Clinical Trials Call Center, Philadelphia, Pennsylvania
- France (2):
  - GSK Clinical Trials Call Center, Lyon
  - GSK Clinical Trials Call Center, Paris
- United Kingdom (2):
  - GSK Clinical Trials Call Center, London
  - GSK Clinical Trials Call Center, Manchester